CLINICAL TRIAL: NCT06809777
Title: Comparison Between the Efficacy and Safety of Topical Podophyllin 25% Versus Cryotherapy in the Treatment of Anogenital Warts
Brief Title: Comparison Between Efficacy of Topical 25%Podophyllin and Cryotherapy on Genital Warts
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Narjis Batool, Post graduate resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SheikhZyMC
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Anogenital Human Papilloma Virus Infection
Keywords: Anogenital warts; Topical 25% podophyllin; cryotherapy
MeSH Terms: conditions — Condylomata Acuminata | interventions — Podophyllin; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 25% podophyllin in treatment of anogenital warts ( Group A ) (Active Comparator): 25% podophyllin resin will be applied topically once weekly for 4 weeks
  Interventions: Drug: Topical 25% podophyllin
- cryotherapy for anogenital warts( Group B) (Active Comparator): cryotherapy of 10 seconds freeze cycle twice weekly for 04 weeks
  Interventions: Procedure: Cryotherapy

INTERVENTIONS:
Drug: Topical 25% podophyllin — 25% podophyllin applied topically once weekly for 4 weeks
  Arms: 25% podophyllin in treatment of anogenital warts ( Group A )
Procedure: Cryotherapy — cryotherapy of 10 sec freeze cycle applied twice weekly for 4 weeks
  Arms: cryotherapy for anogenital warts( Group B)

SUMMARY:
Human papilloma virus (HPV), is the major prevalent cause of sexually transmitted disease affecting genitalia, causing Condylomata Accuminata, also known as external genital warts or anogenital warts.¹ Occurring in men and women with a prevalence rate of 0.6-1.2% worldwide. It primarily affects those in the age range of 20-25 years. Human papilloma virus infections subclinically are primarily caused by either type HPV- 6 or HPV- 11.

A vast variety of treatment options are available to treat CA , including immunomodulators ( imiquimod, purified protein derivative and the HPV vaccine), physical ablation ( cryotherapy and electrodessication) and topical cytotoxic drugs ( TCA, phenol, 5- fluorouracil, retinoids, podophyllin and bleomycin)¹ . Although there are multiple effective treatment are present for EGW, no single treatment has been identified as the best ideal way to treat CA.

Cryotherapy causes the destruction of keratinocytes infected with HPV by using below zero temperature and leading to thermal cell necrosis.

Podophyllum peltatum and Podophyllum emodi are the main source of Podophyllin, a refined plant- based resin.¹² It works by attaching itself to the infected cell's microtubule disturbing the linking process which stops the mitotic process during the metaphase stage of cell division causing the death of epithelial cell.

Study will include patients which will be divided into 2 groups A & B, 48 in each group. Group A will receive topical 25% podophyllin resin via cotton bud under supervision once weekly for 04 weeks. Group B will receive cryotherapy of 10sec freeze cycle twice weekly for 04 weeks. Patient will be followed at interval of 4 weeks and 8 weeks from start of treatment.

Treatment will be considered efficant when decrease in the number of warts is clinically evident at follow up visits. Efficacy of treatment will be graded as 'excellent' >90% clearance, 'good'60-89% clearance, 'satisfactory'30-59% clearance and 'poor'<30% clearance.

DETAILED DESCRIPTION:
Human papilloma virus (HPV), is the major prevalent cause of sexually transmitted disease affecting genitalia, causing Condylomata Accuminata, also known as external genital warts or anogenital warts. Occurring in men and women with a prevalence rate of 0.6-1.2% worldwide. It primarily affects those in the age range of 20-25 years. Human papilloma virus infections subclinically are primarily caused by either type HPV- 6 or HPV- 11.Topical medicines, surgeries and other treatment are among the many possible therapeutic options available. However recurrence and treatment failure are observed with almost all the available treatment after the warts have been visibly cleared.

EGW management poses a major obstacle therapeutically . The patient's immunological condition determine the outcome of the warts , if they are left untreated , they could go away spontaneously, get bigger in size and numerous , or remain the same. The treatment goal is to remove visible warts in order to potentially reduce their infectious , if not the carcinogenic properties.

In this study we will compare the efficacy of topical 25% podophyllin resin versus cryotherapy for the treatment of warts .

Study will include patients which will be divided into 2 groups A & B, 48 in each group. Group A will receive topical 25% podophyllin resin via cotton bud under supervision once weekly for 04 weeks. Group B will receive cryotherapy of 10sec freeze cycle twice weekly for 04 weeks. Patient will be followed at interval of 4 weeks and 8 weeks from start of treatment.

Treatment will be considered efficant when decrease in the number of warts is clinically evident at follow up visits. Efficacy of treatment will be graded as 'excellent' >90% clearance, 'good'60-89% clearance, 'satisfactory'30-59% clearance and 'poor'<30% clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age: 16-60years
* Gender: Any gender
* All new clinically diagnosed cases of plane warts
* Type of warts: plane warts
* Area: Ano-genital warts
* Size: Less than 10cm2(cummulative)
* No. of warts: Upto 20
* Duration of disease: Any

Exclusion Criteria:

* Pregnancy and lactating females
* Bleeding disorders
* Immunocompromised patients.
* Diabetic patients / Peripheral vascular disease.
* Bleeding warts, moles, birthmarks.
* Any other inflammatory dermatosis on that area
* History of any previous treatment in last 2 months.
* Liver/Renal disease
* Hypersensitivity to Podophyllin.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-29 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment will be graded as 'excellent' >90% clearance, 'good'60-89% clearance, 'satisfactory'30-59% clearance and 'poor'<30 | 6 months
  Treatment will be considered efficant when decrease in the number of warts is clinically evident at follow up visits at 4 weeks and 8 weeks after the start of treatment. Efficacy of treatment will be graded as 'excellent' >90% clearance, 'good'60-89% clearance, 'satisfactory'30-59% clearance and 'poor'<30% clearance.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No